CLINICAL TRIAL: NCT01685411
Title: Busulfan and Cyclophosphamide Followed By Allogeneic Hematopoietic Cell Transplantation In Patients With Hematological Malignancies
Brief Title: Busulfan and Cyclophosphamide Followed By ALLO BMT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011OC139; MT2011-20C (Other: Blood and Marrow Transplantation Program)
Record Dates: First submitted 2012-09-05; First posted 2012-09-14 (Estimated); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Allopurinol; Levetiracetam; Busulfan; Cyclophosphamide; Tacrolimus; Mycophenolic Acid; Filgrastim; Granulocyte Colony-Stimulating Factor; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Allogeneic Hematopoietic Stem Cell Transplant (Experimental): Patients treated with Allopurinol, Keppra, Busulfan, Cyclophosphamide, Filgrastim, antithymocyte globulin, Tacrolimus, Mycophenolate mofetil and allogeneic hematopoietic stem cell transplant infusion.
  Interventions: Drug: Allopurinol; Drug: Keppra; Drug: Busulfan; Drug: Cyclophosphamide; Drug: Tacrolimus; Drug: Mycophenolate mofetil; Biological: Allogeneic hematopoietic stem cell transplant; Biological: Filgrastim; Biological: antithymocyte globulin

INTERVENTIONS:
Drug: Allopurinol — Day -8 (prior to transplant): Per institutional guidelines
  Other Names: Lopurin; Zyloprim
Drug: Keppra — Day -8 (prior to transplant): Per institutional guidelines
  Other Names: Levetiracetam
Drug: Busulfan — Days -7 through -4 (prior to transplant): given intravenously (IV) infusion over 2 hours every 6 hours following dose, administration and pharmacokinetic monitoring per University of Minnesota institutional guidelines.
  Other Names: Myleran
Drug: Cyclophosphamide — Days -3 and -2 (prior to transplantation): given as a 2 hour intravenous infusion with a high volume fluid flush and mesna per institutional guidelines. Dosing is based on actual body weight.
  Other Names: Cytoxan
Drug: Tacrolimus — All patients (regardless of allograft source) will receive tacrolimus therapy beginning on day -3. Dosing will be monitored and altered as clinically appropriate per institutional pharmacy guidelines. Dose adjustments will be made on the basis of toxicity and/or low tacrolimus levels. Taper at day +100 for matched sibling donor (MSD) recipients, and day +180 for non-MSD recipients. Taper to zero by 10% weekly dose reduction over approximately 10 weeks.
Drug: Mycophenolate mofetil — Day -3 (prior to transplant): Recipients of umbilical cord blood will given a dose of 3 gm/day every 8 or 12 hours (> or = 40 kg) or 15 mg/kg 3 times per day (< 40 kg) for up to 30 days unless no engraftment.
  Other Names: MMF
Biological: Allogeneic hematopoietic stem cell transplant — Day 0 (or Day+1/+2 to accommodate weekdays): Infusion of cells from related or unrelated donor bone marrow or single or double unrelated donor umbilical cord blood.
Biological: Filgrastim — Beginning Day +1: Intravenously (IV) 5 mcg/kg once daily and continuing until the absolute neutrophil count is >2500 x 10^9/L or per institutional guidelines.
  Other Names: G-CSF; Granulocyte-colony stimulating factor
Biological: antithymocyte globulin — Administered per institutional guidelines for recipients of umbilical cord blood transplant.
  Other Names: ATG

SUMMARY:
This is a treatment guideline to allow routine clinical data to be collected and maintained in Oncore (clinical database) and the University of Minnesota Blood and Marrow Database as part of the historical database maintained by the department.

DETAILED DESCRIPTION:
This is a single arm trial to evaluate the efficacy of busulfan and cyclophosphamide followed by an allogeneic hematopoietic stem cell transplant (HSCT) in the treatment of hematological malignancies. The intent of this study is to provide a protocol that will use unmanipulated allogeneic hematopoietic stem cells from related and unrelated donors after a common preparative regimen.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia (ALL), acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) and current in complete remission meeting one of the following:

  * <45 years of age who are at least 6 months after initial hematopoietic stem cell transplant (HSCT)
  * <45 years of age and have received sufficient radiation treatment to be ineligible for total body irradiation (TBI) containing preparative therapy
* Karnofsky performance status >70% or if <16 years of age, a Lansky play score >50
* Adequate major organ function including:

  * cardiac: left ventricular ejection fraction >45% by echocardiogram (ECHO/MUGA)
  * renal: creatinine clearance >40 mL/min/1.73m^2
  * hepatic: no clinical evidence of hepatic failure (e.g., coagulopathy, ascites)
* An acceptable source of stem cells according to current University of Minnesota Bone Marrow Transplant program guidelines. Acceptable stem cell sources include:

  * HLA-matched related or unrelated donor bone marrow (6/6 or 5/6 antigen match)
  * HLA-matched related or unrelated donor peripheral blood stem cells
  * related or single or double unrelated donor umbilical cord blood (6/6, 5/6 or 4/6 match)
* Women of childbearing age must have a negative pregnancy test and all sexually active participants must agree to use effective contraception during study treatment
* Written consent (adult or parent/guardian)

Exclusion Criteria:

* eligible for TBI containing preparative regimen
* active uncontrolled infection within one week of study enrollment
* pregnant or lactating female

Max Age: 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2013-01; Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret L. MacMillan, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Counts of Participants With Disease Free Survival
Description: The length of time after treatment ends that a patient survives without any signs or symptoms of that cancer or any other type of cancer. In a clinical trial, measuring the disease-free survival is one way to see how well a new treatment works. Patients with leukemia involving the BM and myelodysplastic syndrome will have this assessed by BM biopsy and additional special studies such as cytogenetics or flow cytometry as appropriate. Patients will also have radiology studies such as plain X-rays or CT scans and/or other studies such as blood tumor markers to document presence or absence of disease as clinically indicated.
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
Participants | 3

2. Primary Outcome: Count of Participants With Disease Free Survival
Description: The length of time after treatment ends that a patient survives without any signs or symptoms of that cancer or any other type of cancer. In a clinical trial, measuring the disease-free survival is one way to see how well a new treatment works. Patients with leukemia involving the BM and myelodysplastic syndrome will have this done by BM biopsy and additional special studies such as cytogenetics or flow cytometry as appropriate. Patients will also have radiology studies such as plain X-rays or CT scans and/or other studies such as blood tumor markers to document presence or absence of disease as clinically indicated.
Time Frame: 5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
Participants | 1

3. Primary Outcome: Count of Participants With Disease Free Survival
Description: as for outcome 2
Time Frame: 7 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
Participants | 1

4. Secondary Outcome: Count of Participants Who Achieved Neutrophil Engraftment
Description: Neutrophil engraftment is defined as the first day of three consecutive days where the neutrophil count (absolute neutrophil count) is 500 cells/mm^3 (0.5 x 10^9/L) or greater.
Time Frame: By Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
Participants | 5

5. Secondary Outcome: Percentage of Participants With Acute Graft-Versus-Host Disease by Grade
Description: Acute Graft-Versus-Host Disease is a severe short-term complication created by infusion of donor cells into a foreign host. Patients will be staged weekly between days 0 and 100 after transplantation using standard criteria used for staging. Patients will be assigned an overall GVHD score based on extent of skin rash, volume of diarrhea and maximum bilirubin level. The stages of individual organ involvement are combined to produce an overall grade. Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: Day 100
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
percentage of participants
  Grade 2-4 | 40 [1 to 79]
  Grade 3-4 | 20 [0 to 51]

6. Secondary Outcome: Percentage of Participants With Chronic Graft-Versus-Host Disease
Description: Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cells into a foreign host. Patients will be assigned an overall GVHD score based on extent of skin rash, volume of diarrhea and maximum bilirubin level. The stages of individual organ involvement are combined to produce an overall grade. Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
percentage of participants | 0 [0 to 0]

7. Secondary Outcome: Percentage of Participants With Chronic Graft-Versus-Host Disease
Description: Chronic Graft-Versus-Host Disease is a severe long-term complication created by infusion of donor cells into a foreign host. Patients will be staged weekly between days 0 and 100 after transplantation using standard criteria used for staging. Patients will be assigned an overall GVHD score based on extent of skin rash, volume of diarrhea and maximum bilirubin level. The stages of individual organ involvement are combined to produce an overall grade. Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
percentage of participants | 0 [0 to 0]

8. Secondary Outcome: Percentage of Participants With Treatment-Related Toxicity
Description: In the field of transplantation, toxicity is high and all deaths without previous relapse or progression are usually considered as related to transplantation.
Time Frame: 6 Months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
percentage of participants | 0 [0 to 0]

9. Secondary Outcome: Percentage of Participants With Treatment-Related Toxicity
Description: as for outcome 8
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
percentage of participants | 0 [0 to 0]

10. Secondary Outcome: Percentage of Participants With Relapse
Description: The return of disease after its apparent recovery/cessation. Patients with leukemia involving the BM and myelodysplastic syndrome will have this assessed by BM biopsy and additional special studies such as cytogenetics or flow cytometry as appropriate. Patients will also have radiology studies such as plain X-rays or CT scans and/or other studies such as blood tumor markers to document presence or absence of disease as clinically indicated.
Time Frame: 1 Year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
percentage of participants | 40 [1 to 79]

11. Secondary Outcome: Percentage of Participants With Relapse
Description: as for outcome 10
Time Frame: 2 Years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
percentage of participants | 40 [1 to 79]

12. Secondary Outcome: Percentage of Participants With Engraftment Failure
Description: Graft failure is defined as not accepting donated cells. The donated cells do not make the new white blood cells, red blood cells and platelets.
Time Frame: Day 42
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
percentage of participants | 0 [0 to 0]

13. Secondary Outcome: Number of Participant Who Were Alive at 2 Years Post Transplant
Description: Overall survival will be defined as time from date of enrollment to date of death or censored at the date of last documented contact for patients still alive.
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
Participants | 4

14. Secondary Outcome: Number of Participant Who Were Alive at 5 Years Post Transplant
Description: as for outcome 13
Time Frame: 5 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
Participants | 3

15. Secondary Outcome: Number of Participant Who Were Alive at 7 Years Post Transplant
Description: as for outcome 13
Time Frame: 7 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Time Frame: 7 years
Arm/Group | Allogeneic Hematopoietic Stem Cell Transplant
All-Cause Mortality (participants affected / at risk) | 4/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Allogeneic Hematopoietic Stem Cell Transplant (N=5)
Veno-occlusive disease (VOD) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Bacterial infection (Infections and infestations) | 4 (26)
Brain infarction (Nervous system disorders) | 1 (1)
Cardiac dysfunction (Cardiac disorders) | 1 (1)
Cataracts (Eye disorders) | 1 (1)
CSA induced hypertension (Blood and lymphatic system disorders) | 2 (2)
Engraftment syndrome (General disorders) | 1 (1)
Fungal infection (Infections and infestations) | 1 (3)
GI bleeding (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Intubation (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Multifactorial delirium (Nervous system disorders) | 1 (1)
Neurotoxicity (Nervous system disorders) | 1 (2)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pneumonia (Infections and infestations) | 3 (6)
Renal failure (Renal and urinary disorders) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Transplant-associated thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Viral infection (Infections and infestations) | 2 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-19): https://cdn.clinicaltrials.gov/large-docs/11/NCT01685411/Prot_SAP_000.pdf